CLINICAL TRIAL: NCT05703464
Title: A Multicenter, Single-group, Open-label, Before-and-after Study Confirming Recovery of Defecation Desire by Administration of Elobixibat in Patients With Chronic Constipation
Brief Title: Elobixibat for Chronic Constipation Without Defecation Desire
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Personal reason
Sponsor: International University of Health and Welfare (Other)
Responsible Party: Principal Investigator, Takaomi Kessoku, MD, PhD, International University of Health and Welfare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-Nr-049
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Chronic Constipation
MeSH Terms: interventions — elobixibat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elobixibat (Experimental): 10mg Elobixibat administration for 4 weeks
  Interventions: Drug: Elobixibat 10mg

INTERVENTIONS:
Drug: Elobixibat 10mg — Patients of chronic constipation with loss of defecation desire are administered Elobixibat 10mg for 4 weeks

SUMMARY:
Patients of chronic constipation without defecation desire will be orally administered elobixibat 10 mg once daily before meals for 4 weeks. The primary endpoint of the pre/post comparative study will be the percentage of improvement in bowel movements from Week 2 of the observation period at Week 4 of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

At the time of provisional registration

* Patients diagnosed with chronic constipation using the Rome IV criteria for the diagnosis of chronic constipation
* Age: 20 years or older (at the time of obtaining consent)
* Gender: Any
* outpatients
* Patients for whom written consent can be obtained
* Patients who can record defecation, etc. in the patient diary

At the time of registration ・Dosing start criteria Patients with the following ・'Loss of defecation desire'* in the second week of the observation period (1 week before the start of the treatment period)

*"Loss of defecation desire " refers to patients whose "presence or absence of defecation desire" on the patient questionnaire was "4. almost never" or "5. never".

Exclusion Criteria:

At the time of temporary registration Exclude patients with any of the following conditions

* Patients with organ-related constipation or suspected of having organ-related constipation
* Patients with or suspected of having functional ileus
* Patients with or suspected of having inguinal hernia
* Patients with a history of open abdominal surgery within 12 weeks prior to obtaining consent (excluding appendicitis resection)
* Patients with a history of surgical or endoscopic procedures related to gallbladder resection and papillotomy
* Patients with complications of malignancy However, patients who have undergone radical surgery or who have completed chemotherapy or radiotherapy may be registered.
* Pregnant women, lactating women, women who may be currently pregnant, or patients who cannot give consent to use contraception while participating in the study
* Patients with serious renal, hepatic, or cardiac disease
* Patients with drug allergy to the study drug
* Patients who are participating in other clinical studies, or who have participated in other clinical studies within 4 weeks prior to obtaining consent However, observational studies are excluded.
* Other patients who are judged by the principal investigator or sub-investigator to be inappropriate for this study.

At the time of registration、Dosing start criteria

* Patients who increased the dose of concomitantly restricted drugs during the observation period
* Patients who used concomitantly prohibited drugs during the observation period

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Percentage of change in loss of defecation desire | Week 4
  Percentage of change in loss of defecation desire in the fourth week of the treatment period from the second week of the observation period (patient questionnaire). The presence or absence of defecation desire was assessed using a 5-point scale on the patient questionnaire: 1. always, 2. almost always, 3. a little, 4. almost never, 5. never.

SECONDARY OUTCOMES:
Presence of defecation desire | Week 4
  Changes in the item in each week of the treatment period and comparison of Week 4 of the treatment period with Week 2 of the observation period (patient questionnaire). The presence or absence of defecation desire was assessed using a 5-point scale on the patient questionnaire: 1. always, 2. almost always, 3. a little, 4. almost never, 5. never.
Satisfaction with defecation desire | Week 4
  Changes in the item in each week of the treatment period and comparison of Week 4 of the treatment period with Week 2 of the observation period (patient questionnaire).
Satisfaction of straining | Week 4
  Changes in the item in each week of the treatment period and comparison of Week 4 of the treatment period with Week 2 of the observation period(patient questionnaire).
Degree of straining | Week 4
  Changes in the item in each week of the treatment period and comparison of Week 4 of the treatment period with Week 2 of the observation period(patient questionnaire).
Presence of a sense of incomplete evacuation | Week 4
  Changes in the item in each week of the treatment period and comparison of Week 4 of the treatment period with Week 2 of the observation period (patient questionnaire).
Satisfaction with treatment | Week 4
  Changes in the item in each week of the treatment period and comparison of Week 4 of the treatment period with Week 2 of the observation period (patient questionnaire).
Spontaneous bowel movement (SBM) frequency | Week 4
  Changes in the item in each week of the treatment period and comparison of Week 4 of the treatment period with Week 2 of the observation period (patient daily).
Complete Spontaneous Bowel Movement (CSBM) frequency | Week 4
  Changes in the item in each week of the treatment period and comparison of Week 4 of the treatment period with Week 2 of the observation period (patient daily).
Stool hardness based on the Bristol Stool Form Scale | Week 4
  Changes in the item in each week of the treatment period and comparison of Week 4 of the treatment period with Week 2 of the observation period (patient questionnaire).
Constipation severity score | Week 4
  Comparison of the Constipation severity score at Week 4 of the treatment period with Week 2 of the observation period (patient questionnaire).
Japanese version of the Patient Assessment of Constipation Quality of Life | Week 4
  Comparison of the Japanese version of the Patient Assessment of Constipation Quality of Life questionraire at Week 4 of the treatment period with Week 2 of the observation period (patient questionnaire).
Change of bile acid concentration | Week 4
  Comparison of the bile acid concentration at Week 4 of the treatment period with Week 2 of the observation period (serum and feces).
Change in defecation time. | Week 4
  Changes in the time from taking elobixibat to defecation each week during the treatment period

OTHER OUTCOMES:
Incidence rate of diseases | Week 0-4
  Safety assessment

CONTACTS AND LOCATIONS:
Overall Officials: Takaomi Kessoku, M.D., PhD., Principal Investigator — International university health and welfare Narita hospital
Locations (1):
- International university health and welfare Narita hospital, Narita, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohkubo H, Takatsu T, Yoshihara T, Misawa N, Ashikari K, Fuyuki A, Matsuura T, Higurashi T, Yamamoto K, Matsumoto H, Odaka T, Lembo AJ, Nakajima A. Difference in Defecation Desire Between Patients With and Without Chronic Constipation: A Large-Scale Internet Survey. Clin Transl Gastroenterol. 2020 Sep;11(9):e00230. doi: 10.14309/ctg.0000000000000230. PMID 32858571